CLINICAL TRIAL: NCT01579981
Title: The Exaggerated Glucagon-like Peptide-1 Response is Important for the Improved β-cell Function and Glucose Tolerance After Roux-en-Y Gastric Bypass in Patients With Type 2 Diabetes
Brief Title: The Importance of GLP-1 in Post RYGB Improvement in Glycaemic Control Type 2 Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nils Bruun Jørgensen, Klinisk Assistent, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: H-A-2008-080-31742
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes
Keywords: RYGB; Bariatric Surgery; Glucagon-like-peptide 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — On two separate experimental days before, 1 wk, and 3 months after RYGB, subjects are given a liquid meal test during Exendin 9-39 (900 pmol/min/kg)or saline infusion. The order of the infusions is randomized. At end of study day an ad libitum meal is served.

SUMMARY:
After Roux-en-Y gastric bypass (RYGB) meal induced GLP-1 secretion is dramatically increased, while beta-cell function is increased in type 2 diabetic (T2D) subjects. The aim of this study is to establish causality between the two observations. By meal testing 10 T2D subjects with infusion of saline or exendin (9-39), a GLP-1R specific blocker, before and 1 week and 3 months after RYGB we hope to demonstrate the role of GLP-1 in improveing beta-cell function and maintaing glucose tolerance after RYGB in T2D subjects. Furthermore, effects of GLP-1 rec blockade before and after RYGB on ad libitum energy intake is examined

DETAILED DESCRIPTION:
After Roux-en-Y gastric bypass (RYGB) meal induced GLP-1 secretion is dramatically increased, while beta-cell function is increased in type 2 diabetic (T2D) subjects. The aim of this study is to establish causality between the two observations. By meal testing 10 T2D subjects with infusion of saline or exendin (9-39), a GLP-1R specific blocker, before and 1 week and 3 months after RYGB we hope to demonstrate the role of GLP-1 in improveing beta-cell function and maintaing glucose tolerance after RYGB in T2D subjects. Furthermore, effects of GLP-1 rec blockade before and after RYGB on ad libitum energy intake is examined

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose > 7.0 mM, 2h glucose after OGTT > 11.0 mM. BMI > 35. HbA1c < 8.5%. Fasting C-peptide > 700 pM. Elegible for RYGB.

Exclusion Criteria:

* Dysregulated hypothyroidism, hyperthyroidism, anaemia.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Beta cell glucose sensitivity | 1 week and 3 months after RYGB
  change in prehepatic insulin secretionrate relative to glucose increments

SECONDARY OUTCOMES:
Glucose tolerance | 1 week and 3 months after RYGB
  change in AUC glucose
Ad libitum food intake | 3 months after surgery
  Change in amount of calories ingested

CONTACTS AND LOCATIONS:
Overall Officials: Sten Madsbad, MD, DMSc, Study Chair — Dept. of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark; Nils B Jørgensen, MD, Principal Investigator — Dept. of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark
Locations (1):
- Dept. of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Palleja A, Kashani A, Allin KH, Nielsen T, Zhang C, Li Y, Brach T, Liang S, Feng Q, Jorgensen NB, Bojsen-Moller KN, Dirksen C, Burgdorf KS, Holst JJ, Madsbad S, Wang J, Pedersen O, Hansen T, Arumugam M. Roux-en-Y gastric bypass surgery of morbidly obese patients induces swift and persistent changes of the individual gut microbiota. Genome Med. 2016 Jun 15;8(1):67. doi: 10.1186/s13073-016-0312-1. PMID 27306058
- [Derived] Lindegaard KK, Jorgensen NB, Just R, Heegaard PM, Madsbad S. Effects of Roux-en-Y gastric bypass on fasting and postprandial inflammation-related parameters in obese subjects with normal glucose tolerance and in obese subjects with type 2 diabetes. Diabetol Metab Syndr. 2015 Feb 24;7:12. doi: 10.1186/s13098-015-0012-9. eCollection 2015. PMID 25763111